CLINICAL TRIAL: NCT02381613
Title: Postprandial Plasma Nutrient Differences Between Baked Beef, Baked Herring and Pickled Herring.
Brief Title: Postprandial Differences After Herring and Beef
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Oy Foodfiles Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CSP U-12-001
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Cardiovascular Disease
Keywords: Fish; Herring; Meat; Beef
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baked beef (Active Comparator): A meal based on baked beef
  Interventions: Other: Baked beef
- Baked herring (Experimental): A meal based on baked herring
  Interventions: Other: Baked herring
- Pickled herring (Experimental): A meal based on pickled herring
  Interventions: Other: Pickled herring

INTERVENTIONS:
Other: Baked beef — A meal based on baked beef
  Arms: Baked beef
Other: Baked herring — A meal based on baked herring
  Arms: Baked herring
Other: Pickled herring — A meal based on pickled herring
  Arms: Pickled herring

SUMMARY:
While observational studies often find that diets rich in fish reduce the risk of disease, and that diets including a high intake of red meat are associated with increased risk of cardiovascular disease and cancer, the difference in health effects between red meat and fish are rarely researched in intervention studies.

The investigators hypothesise that the post-prandial plasma response of lipids and markers of cardiovascular disease risk will be more favourable after intake of herring compared to beef.

In addition, while pickling herring in a brine/sugar solution is a common form of preparation, little is known if there is a difference in potential health effects based on the preparation of herring. The investigators will compare baked and pickled herring to understand if preparation is potentially an important factor to be considered when looking at intake of fish and health.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 35-67 years
* BMI >30 kg/m2
* Normally eats lunch and dinner

Exclusion Criteria:

* Smoke or oral tobacco use
* Use of prescription or recreational drugs likely to interfere with primary outcome
* Change in body weight in the month prior to the study
* Abnormal blood biomarker values (assessed by a clinician)

Ages: 35 Years to 67 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Omega-3 fatty acids | Area under the curve between 0 and 7 hours

SECONDARY OUTCOMES:
Plasms insulin | Area under the curve between 0 and 7 hours
Plasma triglycerides | Area under the curve between 0 and 7 hours
Plasma lipoprotein-cholesterol | Area under the curve between 0 and 7 hours
Plasma vitamin D | Area under the curve between 0 and 7 hours
Plasma metabolomic profile | Area under the curve between 0 and 7 hours
Urinary metabolomics | Area under the curve between 0 and 7 hours

REFERENCES:
- [Derived] Ross AB, Svelander C, Undeland I, Pinto R, Sandberg AS. Herring and Beef Meals Lead to Differences in Plasma 2-Aminoadipic Acid, beta-Alanine, 4-Hydroxyproline, Cetoleic Acid, and Docosahexaenoic Acid Concentrations in Overweight Men. J Nutr. 2015 Nov;145(11):2456-63. doi: 10.3945/jn.115.214262. Epub 2015 Sep 23. PMID 26400963